CLINICAL TRIAL: NCT05187949
Title: Promoting Shared-decision Making in Opportunistic Screening for Prostate Cancer
Acronym: PROSHADE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government); Hospital de Sant Pau (Other); Hospital Universitario San Juan de Alicante (Other); Universidad Católica San Antonio de Murcia (Other); Hospital General Universitario de Alicante (Other)
Responsible Party: Principal Investigator, Blanca Juana Lumbreras Lacarra, Professor, Universidad Miguel Hernandez de Elche
Other Study IDs: PI20/01334
Record Dates: First submitted 2021-12-09; First posted 2022-01-12 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Decision Making, Shared; Prostate-Specific Antigen; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients: Quantitative study: Surveys: 1,067 out of a total of 1,389,725 people of residents of the Valencian Community, Spain. Three groups with quota control: proportional to age (40-50; 50-70; > 70 years) of men aged 40 and over who have not had prostate cancer from each stratum (geographical area and population habitat).
  Qualitative study: general population focus groups: 3
  Interventions: Other: Mixed-method approach
- General Practitioners: Quantitative study: 369 General Practitioners working in two Health Departments in the Valencian Community, Spain (Dept of Health Alicante, General Hospital 19, 255,439 habitants) and (Dept of Health Alicante, S Juan Alicante 17, 233,115 habitants).
  Qualitative study: general practitioners focus groups: 2.
  Interventions: Other: Mixed-method approach
- Urologists: Quantitative study: 345 Urologists working in Valencian Community, Spain Qualitative study: urologists focus groups: 1.
  Interventions: Other: Mixed-method approach

INTERVENTIONS:
Other: Mixed-method approach — Quantitative survey (cross-sectional design) and qualitative analysis (focus groups)

SUMMARY:
In this project, the investigators aim to evaluate the most appropriate design and implementation strategy of a decision-aid to promote shared-decision making in prostate cancer screening.

DETAILED DESCRIPTION:
Prostate cancer (PC) screening using Prostate Specific Antigen (PSA) has led to a reduction in advanced disease and disease-specific mortality. However, screening with PSA can also cause harm and is associated with false-positive results and overdiagnosis.

Shared-decision making (SDM) has been defined as the key to successful patient-centered care. The promotion SDM when deciding on PSA screening will have proximal effects such as the development of collaborative deliberation between clinicians and patients, resulting in well-informed patients and in preference-based decisions. As long term effects, it will result in safer, cost-effective, patient-aligned healthcare, and its distant effects will include improvements in resource use, planning processes and improved health outcomes.

The project includes a mixed-method approach. The investigators will perform a quantitative survey (cross-sectional design) to evaluate the population, patients' and clinicians' knowledge about the benefits and risks derived from the PSA determination and the available recommendations.

The investigators will apply qualitative analysis through focus groups, to explore the challenges patients and clinicians face to deep in a prostate screening discussion and to assess the adequacy of different implementation strategies.

The investigators will carry out a user-testing design based on mix-methods (questionnaire and semi-structured review) to evaluate the prototype of the initial decision-aid.

Finally, the investigators will carry out a cluster randomised controlled trial, to assess the results derived from the application of the decision-aid, together with a process evaluation using a combination of both qualitative and quantitative methods to monitor the fidelity of the intervention, the clusters' and patients' response to the intervention as well as the mechanisms of adaptation and change at the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients:

   * Men >40 years old
   * Men who have not had prostate cancer
2. General practitioners:

   * Primary care doctors working in the Valencian Community, Spain.
3. Urologists:

   * Urologists working in the Valencian Community, Spain.

Exclusion Criteria:

1. Patients: None
2. General practitioners: None
3. Urologists: None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Group 1 (patients): Men living in the Valencian Community, Spain. Group 2 (general practitioners): Primary care doctors working in the Valencian Community, Spain.
  Group 3 (urologists): Urologists working in the Valencian Community, Spain.
Sampling Method: Probability Sample
Enrollment: 1781 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Patients' and clinicians' knowledge on PSA test questionnaire developed by the investigators | December 2022
  Quantitative questionnaire to evaluate the target population and clinicians' knowledge about the PSA benefits/risks and the available recommendations. The investigators will develop an ad hoc questionnaire which will be validated through the Delphi Method.
Patients' and clinicians' opinions on PSA test | March 2023
  Focus groups to explore qualitatively the challenge patients and clinicians face when discussing prostate cancer screening and to assess their preferences about different designs and implementation strategies.
Number of patients who participated in a shared-decision making with their clinicians when receiving a PSA test | December 2023
  The investigators will assess the number of patients who participate in a shared- decision making with their clinicians when receiving a PSA test. To assess it, the investigators, through a randomized clinical trial, will apply a new decision-aid developed to a group of patients which will be compared with another group which will have normal care.